CLINICAL TRIAL: NCT01219101
Title: Evaluate the Effect of Ethinyl Estradiol on Polycystic Ovary Syndrome Women Undergoing Intrauterine Insemination
Brief Title: The Effect of Ethinyl Estradiol on Polycystic Ovary Syndrome Women Undergoing Intrauterine Insemination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Royan-Emb-010
Record Dates: First submitted 2010-10-09; First posted 2010-10-13 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2009-03

CONDITIONS: Infertility
Keywords: Ethinyl estradiol; Polycystic ovary syndrome; Intrauterine insemination
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clomiphene citrate and ethinyl estradiol (Experimental): Clomiphene citrate is used in combination of ethinyl estradiol (0.05 mg for 5 days) for induction ovulation of polycystic ovary syndrome women undergoing intrauterine insemination
  Interventions: Drug: clomiphene citrate with ethinyl esteradiol
- clomiphene citrate and placebo (Active Comparator): Clomiphene citrate is used in combination of placebo (for 5 days) for induction ovulation of polycystic ovary syndrome women undergoing intrauterine insemination
  Interventions: Drug: clomiphene citrate with plasebo

INTERVENTIONS:
Drug: clomiphene citrate with ethinyl esteradiol — Clomiphene citrate is used in combination of ethinyl estradiol (0.05 mg for 5 days) for induction ovulation of polycystic ovary syndrome women undergoing intrauterine insemination
  Other Names: Drug Administration
  Arms: clomiphene citrate and ethinyl estradiol
Drug: clomiphene citrate with plasebo — Clomiphene citrate is used in combination of placebo (for 5 days) for induction ovulation of polycystic ovary syndrome women undergoing intrauterine insemination
  Other Names: Drug administration
  Arms: clomiphene citrate and placebo

SUMMARY:
According to the studies CC is successful at inducing ovulation in 50%-75% of cases, but only 30-40% becomes pregnant. The difference has been attributed to a negative action of clomifen citrate(CC) in the form of prolonged antiestrogenic effects on endometrial receptivity. For avoiding of these negative effects, giving ethinyl estradiol in sufficient dosages may be effective. The purpose of this study is comparing pregnancy rates after IUI in women who use CC alone and those who use CC in combination with ethinyl estradiol

DETAILED DESCRIPTION:
The proposal of This study approved by our institutional review boards and institution's ethical committee, and all Participants will sign a written consent before enter to study. All patients will be randomly divided into two groups, A and B. Stimulation will begin on day 3 with the administration of 100 mg of clomifen citrate(CC) daily for 5 days. On day 8, ethinyl estradiol will be given daily for 5 days in group A and placebo will be given for 5 days in group B. Plasma levels of estradiol(E2), Luteinizing hormone (LH) and Follicle-stimulating hormone (FSH) will be evaluated on days 3 and 13 of the menstrual cycle. Ultrasound examination will be done on days 3, 13 and days of HCG administration and IUI for determining of endometrial thickness, number of follicles and size of the dominant follicle.

When the diameter of at least one follicle reached equal or greater than 18 mm, human chronic gonadotrophin (HCG) 10,000 IU will be administered.

The pulsatility index also will be recorded in both uterine arteries on day of HCG administration. A single IUI will be performed 24-36 hours after the administration of hCG. Pregnancy will be confirmed by increasing level of concentration of serum βHCG which will be assessed 14 days after IUI

ELIGIBILITY:
Inclusion Criteria:

* The patients with first treatment cycle
* Age between 25 and 30 years,
* Infertility for at least 2 years' duration,
* Oligomenorrhea or amenorrhea associated with a positive Progesterone challenge test
* Women with normal concentrations of prolactin, free thyroxin and thyroid-stimulating hormone (TSH)

Exclusion Criteria:

* Women whose partners had an abnormal semen analysis according to World Health Organization
* Women who had uterine or tubal abnormalities on hysterosalpingography, and women who had a body mass index of >30 kg/m2.

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy rate | 4-6 weeks after embryos transfer(ET)
  Usage of clomifen citrate on special days can increase pregnancy rate

SECONDARY OUTCOMES:
Duration of stimulation days | 5 days
  usage of clomiphen citrate with ethyl estradiol in patients with poly cystic ovary can stimulate ovulation
Endometrial thickness | 13 days
  effect of using drugs to increase endometrial thickness

CONTACTS AND LOCATIONS:
Overall Officials: hamid gourabi, PhD, Study Chair — President of Royan Institute; Ashraf Moieni, MD, Study Director — Scientific Board
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Moini A, Ahmadi F, Jahangiri N, Ahmadi J, Akhoond MR. A randomized controlled trial evaluating the effect of ethinyl estradiol during clomiphene citrate cycles among women with polycystic ovary syndrome. Int J Gynaecol Obstet. 2015 Nov;131(2):129-32. doi: 10.1016/j.ijgo.2015.06.032. Epub 2015 Sep 8. PMID 26391671
- See also: Royan Institute — http://www.royaninstitute.org